CLINICAL TRIAL: NCT03027817
Title: Cardiac Output and Other Hemodynamic Changes With Prone Position in Cervical Myelopathy Patients Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Dhritiman Chakrabarti (Other)
Responsible Party: Sponsor-Investigator, Dhritiman Chakrabarti, Assistant Professor of Neuroanaesthesiology, National Institute of Mental Health and Neuro Sciences, India
Organization: National Institute of Mental Health and Neuro Sciences, India (Other)
Other Study IDs: NIMHANS
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Hemodynamics Instability
Keywords: Prone positioning; Non-invasive Cardiac Output Monitoring
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prone Positioning — Noninvasive cardiac output monitoring parameters were recorded before and after prone positioning.

SUMMARY:
Positioning a patient in prone position under anaesthesia significantly alters cardiovascular physiology. Cervical myelopathy patients are known to have autonomic dysfunction. Such patients when positioned in prone position under anaesthesia carry a higher risk of developing hemodynamic changes and this can compromise spinal cord perfusion.

This prospective observational study was conducted on 30 patients with cervical myelopathy who underwent surgery in prone position at NIMHANS, Bangalore hospital. The non invasive cardiac output monitor (NICOM, Cheetah Medicals) was used to record various hemodynamic parameters. The hemodynamic parameters were recorded at baseline, post induction, post intubation, prior to prone position, post prone position, and every five minutes thereafter upto 20mins.

The hemodynamic parameters that were recorded using the NICOM monitor:

* HR - Heart rate (beats /min)
* NIBP - non invasive blood pressure (mmHg)
* MAP - mean arterial pressure(mmHg)
* CO - cardiac output (l/min)
* CI - cardiac index (l/min/m2)
* SV - Stroke volume (ml/beat)
* SVV -stroke volume variability (%)
* TPR - total peripheral resistance (dynes. sec/cm5)

ELIGIBILITY:
Inclusion Criteria:

Cervical myelopathy patients undergoing surgery in prone position with:

* ASA Class I , II and III
* Age between 18 to 65 years
* Nurick's grade 2 or more

Exclusion Criteria:

* Atlanto occipital dislocation and cervicomedullary junction pathology
* Tumour pathology
* Diabetic patients
* Patients positioned prone in the awake state (without induction of anaesthesia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cervical Myelopathy undergoing elective cervical decompression in prone position.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in mean arterial pressure at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.

SECONDARY OUTCOMES:
Heart rate | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in heart rate at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.
Cardiac output | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in cardiac output at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.
Stroke volume | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in stroke volume at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.
Stroke volume variation | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in stroke volume variation at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.
Total peripheral resistance | Before induction of anaesthesia to 20 minutes after prone positioning (end of study)
  Analysis of change in total peripheral resistance at following time points - before induction of anaesthesia, 2 minutes after anaesthetic induction, 2 minutes after intubation, before turning prone, immediately after turning prone and every 5 minutes thereafter till 20 minutes after positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Manohar, MD, DNB, DM, Principal Investigator — National Institute of Mental Health and Neuro Sciences, Bangalore

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers. If required, the Sponsor-Investigator may be contacted via email shared on this portal.